CLINICAL TRIAL: NCT04405453
Title: Contribution of Erector Spina Plane Block to Analgesia Combined With Ultrasound Guided Trapezius Muscle Injection for Myofascial Pain Syndrome
Brief Title: Contribution of Erector Spina Plane Block to Analgesia for Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, MD, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: DiskapiTRH Algology
Record Dates: First submitted 2020-05-19; First posted 2020-05-28 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Trigger Point; Myofascial Pain
Keywords: Trigger point , Erector spinae plane block , Ultrasonography

STUDY DESIGN:
Intervention Model Description: Patients with myofasial pain syndrome will randomized into two group. TMI group will receive ultrasound guided trapezius muscle injection two times with one week interval. ESPB group in the 1th week will receive ultrasound guided trapezius muscle injection and in the 2nd week ultrasound guided erector spina plane block will receive. Pain severity of the patients will evaluate by visual analog scale. Datas will obtaine before (week 0) and after (week 1,2,3,4) the injections.
Who Masked: Investigator
Masking Description: One physician who will be blind will examinade all patients for eligibility and will valuate the outcome measures although the physician who will performe all injections will not be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trapezius Muscle İnjection (TMI) group (Active Comparator): TMI group will receive ultrasound guided trapezius muscle injection two times with one week interval. Pain severity of the patients will evaluate by visual analog scale before (week 0) and after (week 1,2,3,4) the injections
  Interventions: Procedure: trapezius muscle injection
- Erector Spina Plane Block (ESPB) group (Active Comparator): ESPB group in the 1th week will receive ultrasound guided trapezius muscle injection and in the 2nd week ultrasound guided erector spina plane block will receive. Pain severity of the patients will evaluate by visual analog scale before (week 0) and after (week 1,2,3,4) the injections
  Interventions: Procedure: trapezius muscle injection; Procedure: erector spina plane block

INTERVENTIONS:
Procedure: trapezius muscle injection — TMI group will receive ultrasound guided trapezius muscle injection two times with one week interval.
Procedure: erector spina plane block — 1th week will receive ultrasound guided trapezius muscle injection and in the 2nd week ultrasound guided erector spina plane block will receive
  Arms: Erector Spina Plane Block (ESPB) group

SUMMARY:
Myofascial pain syndrome is a common chronic disease characterized by pain and tenderness in one or more muscle groups. It is characterized by myofascial trigger points that are felt as a band or a nodule harder than normal consistency located in the muscle. Myofascial trigger points are developes as a result of muscle injury ; this can be acute trauma caused by sport injury, accident, or chronic muscle overuse by repetitive occupational activities, emotional stress or poor posture. Trigger point injection is the application of low dose local anesthetic drug into the trigger point.Its main purpose is to weaken the trigger point caused by muscle spasm.However, it may reduce pain partially or have a short duration of action, so it may need to be repeated several times at regular intervals.Trigger point injection can reach trigger points in superficial muscles With the erector spina plane block technique, more effective and long-term pain treatment can be achieved by reaching deeper trigger points. With this hypothesis, we aimed to investigate the contribution of the erector spina plane block to trigger point injection in the treatment of myofascial pain.

DETAILED DESCRIPTION:
Myofascial pain syndrome is a common chronic disease characterized by pain and tenderness in one or more muscle groups. It is characterized by myofascial trigger points that are felt as a band or a nodule harder than normal consistency located in the muscle. Myofascial trigger points are developes as a result of muscle injury ; this can be acute trauma caused by sport injury, accident, or chronic muscle overuse by repetitive occupational activities, emotional stress or poor posture. Trigger point injection is the application of low dose local anesthetic drug into the trigger point.Its main purpose is to weaken the trigger point caused by muscle spasm.However, it may reduce pain partially or have a short duration of action, so it may need to be repeated several times at regular intervals.Trigger point injection can reach trigger points in superficial muscles With the erector spina plane block technique, more effective and long-term pain treatment can be achieved by reaching deeper trigger points. With this hypothesis, we aimed to investigate the contribution of the erector spina plane block to trigger point injection in the treatment of myofascial pain.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Myofascial pain

Exclusion Criteria:

Cervical radiculopathy fibromyalgia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-05 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
VAS (visual analog scale ) score | before injection (week 0)
  Severity of pain The patient rated pain on a scale of 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable.
VAS (visual analog scale ) score | 1st week after injection
  Severity of pain The patient rated pain on a scale of 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable.
VAS (visual analog scale ) score | 2nd week after injection
  Severity of pain The patient rated pain on a scale of 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable.
VAS (visual analog scale ) score | 3rd week after injection
  Severity of pain The patient rated pain on a scale of 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable.
VAS (visual analog scale ) score | 4th weeks after injection
  Severity of pain The patient rated pain on a scale of 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: damla yürük, Principal Investigator — Diskapi Teaching and Research Hospital; ömer taylan akkaya, Study Director — Diskapi Teaching and Research Hospital; Hüseyin Alp Alptekin, Study Chair — Diskapi Teaching and Research Hospital
Locations (1):
- Dişkapi Reserch and Education Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 19.05.2020
Access Criteria: NO CRİTERİA